CLINICAL TRIAL: NCT06853483
Title: School-EduSmoke: A Cluster Randomized Controlled Trial for Promoting Smoking Cessation Among Parents of Schoolchildren
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yanhong Gong, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: S133
Record Dates: First submitted 2025-02-23; First posted 2025-03-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Students in control group will have regular health education classes . Parents in control group will not receive any intervention other than completion questionnaires and cotinine testing.
- Intervention group (Experimental): Students and parents of smokers in the intervention group will work together to receive home-school based smoking cessation intervention strategies.
  Interventions: Behavioral: Family-School based smoking cessation intervention package

INTERVENTIONS:
Behavioral: Family-School based smoking cessation intervention package — The Family-School based smoking cessation intervention programme will be developed using the multiple strategies provided by the BCW framework, with face-to-face + online as the primary mode of implementation. Specifically, educational training based on the school curriculum will be conducted to create a supportive environment for smokers to quit, guide smokers to discover motivation to quit, encourage smokers to cope with key barriers to quitting, as well as incorporate relapse prevention strategies, using formats such as online videos and supplemental materials, with interventions designed to help students and parents of smokers to understand the health hazards of smoking, to enhance cessation action and supportive skills, and inspire healthy action.
  Arms: Intervention group

SUMMARY:
This study is a pragmatic two-group, multi-center, randomized controlled superiority trial, including an internal pilot, economic evaluation and process evaluation, aiming to assess the impact of a school-based comprehensive intervention on smoking cessation actions among parents who smoke.

DETAILED DESCRIPTION:
The School-EduSmoke project will be based on the Behavior change wheel (BCW) and theoretical domain framework. The goal of our project is to promote smoking cessation actions by parents through smoking cessation education for children and their parents in schools. The programme will enhance the implementation of smoking cessation behaviours by identifying key risk factors that influence smoking behaviour, helping to design specific interventions that will particularly help to address ambivalence and defensiveness among smokers. A set of randomized controlled trials will be used to evaluate the effectiveness of the intervention. The findings will provide evidence and support for the provision of low-cost, low-resource, widely accessible smoking cessation support to the smoking community, thereby promoting the effective implementation of smoke-free health actions.

ELIGIBILITY:
Inclusion Criteria:

1. Primary 4 students and their smoking parents.
2. The student has a parent who is a smoker (a smoker is defined as smoking at least 1 cigarette per day).
3. The student and participating parent reside together on a long-term basis.
4. The student and parents have the cognitive, understanding and communication skills to voluntarily participate in this project.

Exclusion Criteria:

* 1) The parent who smokes is currently using other tobacco substances, has recently participated in nicotine replacement therapy, or has other substance abuse.

  2) The parent or student has a serious organic or somatic disease. 3) The parent or student is unwilling to cooperate with the test or refuses to answer questions.

  4) The parent or student has a serious illness that is life-threatening or requires regular hospitalisation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-05-03 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated 24-hour point smoking cessation rate at 6 month | 6-month followup
  Assessing smoking cessation in parents by measuring their urine cotinine levels

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence quit rate | 6 month follow-up
  Subjects reporting not smoking in the past 7-days at 6-month will be regarded asabstinence from smoking. The self-reported 7-days prevalence quit rate will be assessedat the baseline and 6-month later after the intervention.
  "Have you smoked a cigarette (even a puff) in the past 7 days?""
50% reduction in the number of cigarettes smoked | 6-month follow-up
  Cigarette consumption reduced by at least 50% compared with the baseline, the cigarette consumption will be assessed at the baseline and 6-month late after the intervention. "How many cigarettes do you smoke on average per day?"
The level of readiness to quit | 1-month and 6-month follow-up
  "When do you plan to start quitting smoking?" The readiness to quit is divided into pre-contemplation stage (attempt to quitmore that 30 days later), contemplation stage (attempt to quit within 30 daysbut more than 7 days), preparation stage (attempt to quit within 7 days), andaction stage (quitting).

CONTACTS AND LOCATIONS:
Locations (1):
- Dongxihu Primary School, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No